CLINICAL TRIAL: NCT05227560
Title: The Effect of the Emotional Freedom Technique on Students' Anxiety and Coping Styles With Stress During the COVİD-19 Pandemic
Brief Title: The Effect of the Emotional Freedom Technique on Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Canan Eraydın, Lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ZngldkBEU
Record Dates: First submitted 2021-12-29; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Coping Skills; Anxiety; Complementary Therapies; Stress
MeSH Terms: conditions — Anxiety Disorders | interventions — Complementary Therapies

STUDY DESIGN:
Intervention Model Description: This study was carried out in an experimental design with pretest-posttest control group in order to determine the effect of Emotional Freedom Technique (EFT) application on nursing students' anxiety and stress coping styles during the COVID-19 pandemic.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Freedom Technique group (Experimental): Personal characteristics questionnaire, State Anxiety Scale (SQS) and Stress Coping Styles Scale (SST) were applied to the intervention group at the pre-test stage. Subjective discomfort level scale (ERDS) was also applied to the intervention group before EFT was applied. After four sessions of EFT, "DKO", "SBO", "ORDS" were applied to the intervention group again in the post-test phase.
  Interventions: Other: Complementary Therapies
- Control (No Intervention): Participants in the control group received no intervention throughout the study.

INTERVENTIONS:
Other: Complementary Therapies — The emotional freedom technique was applied to the experimental group.
  Arms: Emotional Freedom Technique group

SUMMARY:
Introduction: The interruption of education within the scope of quarantine and isolation methods during the pandemic process has caused nursing students studying in clinical practice areas to be away from the clinic for a long time. This situation not only affected the anxiety levels of nursing students, but also caused them to feel inadequate and to experience stress.

Purpose: The aim of this study is to investigate the effect of emotional freedom technique on nursing students' styles of coping with anxiety and stress.

Method:In this experimentally designed study with pretest-posttest control group, freedom of emotion technique will be applied to the experimental group for 4 sessions. In the pre-implementation phase and after the emotional freedom technique session, the state anxiety scale, coping styles scale, and subjective discomfort level scale will be applied.

DETAILED DESCRIPTION:
Emotional Freedom Technique (EFT), a type of energy that has been applied recently, is a technique applied by touching meridian points to provide anxiety, depression, burnout, stress management, and desensitization to fear. The basic principle of EFT is to send activation and deactivation signals to the brain by stimulating points on the skin with different electrical properties, usually by touching them. The findings obtained from the studies show that this technique, which is a psychotherapeutic technique and provides cognitive restructuring, has statistically significant improvements at the rate of 98% in the management of psychological problems. Studies show that this approach is positive in coping with stress when considered in a wide range. Church et al. revealed that self-administered EFT provides significant improvements in anxiety, depression, pain and craving scores. A large therapeutic effect for EFT was reported in a meta-analysis of 14 randomized controlled trials using the EFT technique for anxiety disorders. In the studies, it was aimed to apply this application, which has proven positive results, to apply the emotional freedom technique in order to reduce the anxiety experienced by the students due to the reasons such as distance education and clinical education during the COVID-19 pandemic process and to enable them to cope with stress.

research questions

This study aims to address the following research questions:

What are the anxiety levels of the students who applied the emotional freedom technique (EFT)? What are the stress coping styles of the students who applied emotional freedom technique (EFT)?

ELIGIBILITY:
Inclusion criteria:

* Not receiving any psychiatric diagnosis,
* Not receiving any therapy for coping with anxiety and stress,
* Not applying emotional freedom technique before,
* Not being in the COVID-19 diagnosis, treatment care process, and
* Participating in the study determined to be voluntary.

Exclusion Criteria:

-Not participating in any of the EFT sessions and being diagnosed with COVID-19.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | 4 months
  State-Trait Anxiety Inventory (STAI) was developed by Spielberger et al. in 1970. It was adapted to Turkish society in 1985 by Öner and Le Compte. The STAI is a scale that separately measures state and trait anxiety levels, with 20 items scored by a Likert scale. The expressions in the scale range from "rarely" to "almost always ."There are two types of expressions in the State-Trait Anxiety scales. Direct expressions express negative feelings, and inverted expressions express positive feelings. Reversed expressions in the state anxiety scale (SAS) are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. Reversed expressions in the trait anxiety scale (TAS) are 21, 26, 27, 30, 33, 36, and 39. The total score obtained from both scales varies between 20 and 80. High scores indicate a severe form of anxiety, whereas low scores indicate a mild form of anxiety
Ways of Coping with Stress Inventory (WCI) | 4 months
  The ways of coping with stress inventory (Appendix 5) was developed by Şahin and Durak (1995) based on the Ways of Coping Inventory developed by Folkman and Lazarus (1984) in order to measure the level of coping skills with stress. The 30-item scale has five sub-dimensions: Self-Confident, Optimistic, Submissive, Helpless styles, and Seeking Social Support. The averages obtained by dividing the scores obtained by the number of questions give information about the coping strategy levels. For example, a score between 0-3 can be obtained from a sub-dimension. While self-confident, optimistic, and seeking social support are active coping strategies, the self-blaming, and submissive approach is one of the passive coping strategies
The subjective units of distress scale (SUD) | 4 months
  The cognitive element of EFT involves self-rating of distress severity and pairing of an abbreviated exposure statement and a self-acceptance statement. The severity of distress is evaluated by subjects on an 11- point Likert scale. 0 corresponds to absolutely no distress, while ten corresponds to the maximum possible distress. This situation is considered as the subjective units of distress scale (SUD) and provides clinicians and patients with the measurement of the severity of symptoms experienced by the latter in addition to a repeated measure by which the progress of treatment can be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Canan Eraydın, Doctorate, Study Director — Bülent Ecevit University
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months